CLINICAL TRIAL: NCT04117347
Title: Morning Light Treatment for Traumatic Stress: The Role of Amygdala Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00161267; 1R61MH117157-01A1 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stress
Keywords: Circadian timing; Mood; Light

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to study arm. The PI, study coordinator and research assistants will remain unblinded to perform safety assessments and provide feedback on intervention adherence. Blinded staff will wear buttons as an upfront visual cue to remind participants not to talk about their treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Light therapy A via the Re-Timer® (Experimental): -15 minutes/day
  Interventions: Device: Light therapy A via the Re-Timer®
- Light therapy B via the Re-Timer® (Experimental): -30 minutes/day
  Interventions: Device: Light therapy B via the Re-Timer®
- Light therapy C via the Re-Timer® (Experimental): -60 minutes/day
  Interventions: Device: Light therapy C via the Re-Timer®

INTERVENTIONS:
Device: Light therapy A via the Re-Timer® — Subjects will conduct light treatment in the mornings at home.
  Other Names: Re-Timer®
  Arms: Light therapy A via the Re-Timer®
Device: Light therapy B via the Re-Timer® — Subjects will conduct light treatment in the mornings at home.
  Other Names: Re-Timer®
  Arms: Light therapy B via the Re-Timer®
Device: Light therapy C via the Re-Timer® — Subjects will conduct light treatment in the mornings at home.
  Other Names: Re-Timer®
  Arms: Light therapy C via the Re-Timer®

SUMMARY:
The purpose of this study is to determine the effect of different amounts of time of morning light on brain emotional processing.

DETAILED DESCRIPTION:
Brain emotional processing was determined with the Emotional Faces Assessment Task (EFAT). In this task, participants view a trio of faces and match one of the two faces (bottom) that expresses the same emotion as the target face (top). The faces display one of five expressions (angry, happy, fearful, sad, neutral) and the other (incongruent) probe face always displays a neutral (or happy if the target is neutral) expression. The paradigm consists of 20 face trials per expression and 20 shape trials, presented in pseudorandomized order, separated by a 3-7 sec intertrial blank screen with fixation cross.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for traumatic stress
* Normal or corrected to normal vision
* Right-handed
* Fluency in English
* Physically able to travel for study visit attendance

Exclusion Criteria:

* Significant chronic uncontrolled disease (e.g. uncontrolled diabetes, advanced liver disease, cancer, etc.)
* Severe hearing problem
* Intellectual disability or serious cognitive impairment
* Inability to tolerate enclosed spaces (e.g. the MRI machine)
* Ferrous-containing metals within the body
* Pregnant, trying to get pregnant, or breastfeeding
* Epilepsy
* Other research participation
* Frequent number of special events during study period (weddings, concerts, exams, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burgess, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are open to sharing data by any appropriate mechanism indicated by NIH program staff. That includes that identified research information will be entered into the National Institute of Mental Health's Database for Clinical Trials related to Mental Illness (NDCT)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After scientific papers are accepted for publication and the data will be available for 7 years after study completion.
Access Criteria: Researchers requesting data will first have to sign a data sharing agreement, agreeing to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, electronically securing the data while in use, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, no use of the data for commercial purposes and proper acknowledgement of the data resource.

REFERENCES:
- [Result] Burgess HJ, Rizvydeen M, Huizenga B, Prasad M, Bahl S, Duval ER, Kim HM, Phan KL, Liberzon I, Abelson J, Klumpp H, Horwitz A, Mooney A, Raglan GB, Zalta AK. A 4-week morning light treatment reduces amygdala reactivity and clinical symptoms in adults with traumatic stress. Psychiatry Res. 2024 Dec;342:116209. doi: 10.1016/j.psychres.2024.116209. Epub 2024 Sep 21. PMID 39316998
- See also: doi — https://doi.org/10.1016/j.psychres.2024.116209

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants withdrew after study enrollment but before randomization.
Groups:
- Light Therapy A Via the Re-Timer®: -15 minutes/day
  Light therapy A via the Re-Timer®: Subjects conducted light treatment in the mornings at home.
- Light Therapy B Via the Re-Timer®: -30 minutes/day
  Light therapy B via the Re-Timer®: Subjects conducted light treatment in the mornings at home.
- Light Therapy C Via the Re-Timer®: -60 minutes/day
  Light therapy C via the Re-Timer®: Subjects conducted light treatment in the mornings at home.
Period: Overall Study
Arm/Group | Light Therapy A Via the Re-Timer® | Light Therapy B Via the Re-Timer® | Light Therapy C Via the Re-Timer®
Started | 15 | 15 | 16
Completed | 14 | 13 | 15
Not Completed | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — No time for study | 0 | 2 | 0
Not completed — Family emergency | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Therapy A Via the Re-Timer® | Light Therapy B Via the Re-Timer® | Light Therapy C Via the Re-Timer® | Total
Number analyzed (Participants) | 15 | 15 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.10 (12.03) | 36.45 (10.58) | 30.69 (8.85) | 33.68 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 34
  Male | 3 | 3 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 14 | 13 | 15 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 12 | 12 | 13 | 37
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 16 | 46
fMRI BOLD signal change in amygdala [Mean (Standard Deviation); unit: beta weight] — Participants completed the Emotional Faces Assessment Task (EFAT) during the fMRI scan. The average blood-oxygen-level-dependent (BOLD) signal change between the display of negative faces versus display of shapes was derived for the left and right amygdala separately. Population: Data from some participants were lost due to poor task performance in the fMRI. This included 0 participants in the Light Therapy A group (15 minute), 1 participant in the Light Therapy B group (30 minute) and 2 participants in the Light Therapy C group (60 minute).
  beta weight
    fMRI BOLD signal change in left amygdala: number analyzed (Participants) | 15 | 14 | 14 | 43
    fMRI BOLD signal change in left amygdala | 0.1311 (0.0816) | 0.1410 (0.0822) | 0.2065 (0.1333) | 0.1589 (0.1047)
    fMRI BOLD signal change in right amygdala: number analyzed (Participants) | 15 | 14 | 14 | 43
    fMRI BOLD signal change in right amygdala | 0.1611 (0.1577) | 0.1800 (0.0936) | 0.1858 (0.0812) | 0.1753 (0.1147)

OUTCOME MEASURES:

1. Primary Outcome: Change in Amygdala Reactivity as Measured by Blood-oxygen-level-dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Signal
Description: Participants completed the Emotional Faces Assessment Task (EFAT) during the fMRI scan. The average blood-oxygen-level-dependent (BOLD) signal change between the display of negative faces versus display of shapes was derived for the left and right amygdala separately. Higher levels indicate greater amygdala reactivity to negative faces versus display of shapes.
Time Frame: Baseline and treatment week 2 and treatment week 4
Population: Four participants discontinued the study after randomization: 2 no time for study (Light Therapy B group -30 minute), 1 family emergency (Light Therapy A group - 15 minute), 1 light-triggered headaches (Light Therapy C group - 60 minute). Some participants were not scanned at week 2 due to various reasons (e.g. weather, available funding).
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Light Therapy A Via the Re-Timer® | Light Therapy B Via the Re-Timer® | Light Therapy C Via the Re-Timer®
Number analyzed (Participants) | 14 | 12 | 13
beta weights
  Baseline (left amygdala) | 0.1287 (0.0842) | 0.1532 (0.0828) | 0.2134 (0.1362)
  After 2 weeks of light treatment (left amygdala): number analyzed (Participants) | 10 | 8 | 8
  After 2 weeks of light treatment (left amygdala) | 0.1048 (0.0770) | 0.1248 (0.0855) | 0.0806 (0.1582)
  After 4 weeks of light treatment (left amygdala) | 0.1155 (0.0927) | 0.1191 (0.1047) | 0.1375 (0.1399)
  Baseline (right amygdala) | 0.1437 (0.1480) | 0.1969 (0.0882) | 0.1899 (0.0830)
  After 2 weeks of light treatment (right amygdala): number analyzed (Participants) | 10 | 8 | 8
  After 2 weeks of light treatment (right amygdala) | 0.1104 (0.0715) | 0.1176 (0.1042) | 0.1012 (0.0716)
  After 4 weeks of light treatment (right amygdala) | 0.1087 (0.1159) | 0.1107 (0.1141) | 0.1303 (0.0905)
Statistical Analysis 1: Comparison: Light Therapy A Via the Re-Timer® vs Light Therapy B Via the Re-Timer®; Analysis for left amygdala; Test type: Other — Dose Response Relationship; Coefficient for an indicator = 0.022, 95% CI 2-sided [-0.0861723 to 0.1309519], Standard Error of Mean 0.054 — coefficient for an indicator for Light Therapy B (vs. Light Therapy A)
Statistical Analysis 2: Comparison: Light Therapy A Via the Re-Timer® vs Light Therapy C Via the Re-Timer®; Analysis for left amygdala; Test type: Other — Dose Response Relationship; Coefficient for an indicator = 0.068, 95% CI 2-sided [-0.0363877 to 0.1730965], Standard Error of Mean 0.052 — coefficient for an indicator for Light Therapy C (vs. Light Therapy A)
Statistical Analysis 3: Comparison: Light Therapy A Via the Re-Timer® vs Light Therapy B Via the Re-Timer®; Analysis for right amygdala; Test type: Other — Dose Response Relationship; Coefficient for an indicator = 0.043, 95% CI 2-sided [-0.0676154 to 0.1545869], Standard Error of Mean 0.055 — coefficient for an indicator for Light Therapy B (vs. Light Therapy A)
Statistical Analysis 4: Comparison: Light Therapy A Via the Re-Timer® vs Light Therapy C Via the Re-Timer®; Analysis for right amygdala; Test type: Other — Dose Response Relationship; Coefficient for an indicator = 0.018, 95% CI 2-sided [-0.0888691 to 0.1255146], Standard Error of Mean 0.053 — coefficient for an indicator for Light Therapy C (vs. Light Therapy A)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Light Therapy A Via the Re-Timer® | Light Therapy B Via the Re-Timer® | Light Therapy C Via the Re-Timer®
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Light Therapy A Via the Re-Timer® (N=15) | Light Therapy B Via the Re-Timer® (N=15) | Light Therapy C Via the Re-Timer® (N=16)
Light-triggered headache (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT04117347/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT04117347/ICF_000.pdf